CLINICAL TRIAL: NCT04300972
Title: Comparison of Contrast Agent Administration Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Kristian Fosså, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CMProtokoll
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Radiography, Thoracic
Keywords: computed tomography; contrast dose; weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixed dose (Other)
  Interventions: Diagnostic Test: Standard dose
- weight and body type adapted dose (Experimental)
  Interventions: Diagnostic Test: Body/weight adaption

INTERVENTIONS:
Diagnostic Test: Body/weight adaption — contrast media dose is adapted to weight and body type
  Arms: weight and body type adapted dose
Diagnostic Test: Standard dose — a fixed amount of contrast media is used, independently of weight and body type
  Arms: fixed dose

SUMMARY:
The will compare two different ways of administering contrast media in CT exams of the chest:

1. a fixed dose of contrast medium
2. a weight- and body-type-adapted dose of contrast medium

The goal is to see if one protocol is superior to the other in reliably producing diagnostic CT images.

DETAILED DESCRIPTION:
The continuing advances in computed tomographic (CT) technology in the past decades have provided ongoing opportunities to improve CT image quality, clinical practice and discover new clinical CT imaging applications. New CT technology, however, has introduced new challenges in clinical radiology practice. One of the challenges deals with intravenous contrast medium (CM) administration. Although multidetector CT allows more efficient and flexible use of contrast medium than single-detector CT, to fully reap the benefits of multidetector CT, certain technical challenges involving maximum contrast enhancement and optimal contrast material delivery must be met (1). While CT technology has evolved, the practice of CT intravenous CM administration has been continually debated and updated. The users of new CT technology, accompanied with its newly added technical complexity, discover they fall short of achieving a desired image quality with the traditional standard administration of CM. This entails a change in practice. In the department of Radiology at St Olav University Hospital (SOH), a new protocol for CM administration is now developed and is ready for implementation. This protocol is based on a body weight adapted CM administration, while the current protocol has a fixed CM injection. In this study, this newly CM administration protocol for thoracic CT will be compared to the fixed CM injection protocol. To our knowledge, very few studies (2) have been published on the use of body weight adapted injection protocols for Thoracic CT. Most of the studies report the impact of body weight adapted CM injection protocols for the coronary arteries of CT angiography (3- 5). Therefore, the aim of this study is to determine whether individually tailored protocol(s) for the injection of CM results in higher and more homogeneous vascular attenuation at thoracic CT compared with conventional injection protocols using fixed injection parameters. We know that to achieve optimal contrast enhancement in thoracic CT involves essential factors such as CT tube voltage and CT attenuation, patient factors, CM factors and CT scanning factors (1) and thus all these factors will be addressed and discussed in this investigation.

Specific aims of the study:

1. To assess and compare the CT attenuation achieved with both protocols
2. Compare the required amount of CM using weight adapted CM protocol and fixed CM injection protocol
3. Compare the quality of the images using weight adapted CM protocol and fixed CM injection protocol

ELIGIBILITY:
All patients referred for a thoracic CT (only) at St. Olavs Hospital will be screened for eligibility Inclusion criteria are

-referral indicates the need for contrast administration (as decided by a radiologist)

Exclusion criteria are:

* impaired renal function (glomerular filtration rate <60 ml/min)
* congenital heart disease (as indicated by referral)
* congestive heart failure (as indicated by referral)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
CT density of large vessel, measured in Hounsfield units (HU) in the imaging software (PACS) | immediately after imaging

IPD SHARING:
Plan to Share IPD: Undecided